CLINICAL TRIAL: NCT02209493
Title: The Efficacy of Nopales (Opuntia Spp.) on Lipoprotein Profile and Oxidative Stress Among Moderately Hypercholesterolemic Adults
Brief Title: Effects of Nopales (Opuntia Spp.) on Lipoprotein Profile and Oxidative Stress in Moderately Hypercholesterolemic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Sonia Vega-Lopez, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Nopales-2014
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Disease
Keywords: Dietary intervention; Hypercholesterolemic adults; Vegetable intake; Functional food; Prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Food supplementation: nopales (Experimental): Consumption of 2 cups/day of cooked nopales (prickly pear cactus leaves) with each of two main meals for 2 weeks
  Interventions: Behavioral: Food supplementation: nopales
- Food supplementation: cucumber (Sham Comparator): Consumption of 2 cups/day peeled and chopped cucumber with each of two main meals for 2 weeks
  Interventions: Behavioral: Food supplementation: cucumber

INTERVENTIONS:
Behavioral: Food supplementation: nopales — Consumption of 2 cups/day of test food: nopales
  Arms: Food supplementation: nopales
Behavioral: Food supplementation: cucumber — Consumption of 2 cups/day of test food: cucumber
  Arms: Food supplementation: cucumber

SUMMARY:
In light of the high CVD morbidity and mortality, promoting simple interventions to improve serum lipids and decrease oxidative stress are warranted to help prevent chronic diseases. Because of their fiber content, nopales (prickly pear cactus pads from the Opuntia species) are commonly regarded among Mexicans as a medicinal plant for glycemic and cholesterol control. However, the literature documenting their purported hypocholesterolemic potential is scarce. Given the unique composition and potential benefits of nopales, their use may be an ideal approach as an adjunct therapy for the reduction in cardiometabolic risk factors. Therefore, the aim of this study is to evaluate the efficacy of a 2-week intervention with nopales pads for the reduction of established CVD risk factors (serum lipids) in comparison to a control food with lower antioxidant and fiber content (cucumber) among adults with moderate hypercholesterolemia in a randomized controlled crossover trial. Because limited data exists on the effects of nopales supplementation on other factors associated with cardiometabolic risk, an exploratory assessment of how biomarkers of insulin sensitivity, inflammation (high sensitivity C-reactive protein [hsCRP]) and oxidative stress (LDL oxidizability and total antioxidant capacity) will also be conducted.

DETAILED DESCRIPTION:
In light of the high cardiovascular disease morbidity and mortality, promoting simple interventions to improve serum lipids and decrease oxidative stress are warranted to help prevent chronic diseases. Commonly prescribed dietary interventions for cardiovascular disease risk reduction include the use of functional foods known to have beneficial effects on risk factors.

Because of their fiber content, nopales (prickly pear cactus pads from the Opuntia species) are commonly regarded among Mexicans as a medicinal plant for glycemic and cholesterol control. However, the literature documenting their purported hypocholesterolemic potential is scarce. Most studies have focused on the prickly pear fruit, rather than the actual nopales cactus pads. Given the unique composition and potential benefits of nopales, their use may be an ideal approach as an adjunct therapy for the reduction in cardiometabolic risk factors.

The aim of this study is to evaluate the efficacy of a 2-week intervention with nopales pads for the reduction of established CVD risk factors (serum lipids) in comparison to a control food with lower antioxidant and fiber content (cucumber) among adults with moderate hypercholesterolemia in a randomized controlled crossover trial. Because limited data exists on the effects of nopales supplementation on other factors associated with cardiometabolic risk, an exploratory assessment of how biomarkers of insulin sensitivity, inflammation (high sensitivity C-reactive protein [hsCRP]) and oxidative stress (LDL oxidizability and total antioxidant capacity) will also be conducted.

In this randomized crossover trial, healthy adults with moderate hypercholesterolemia (LDL-cholesterol ≥ 120 mg/dL) but otherwise healthy will be randomly assigned to supplementation with 2 cups/day of nopales (300 g; intervention) or cucumbers (208 g; control), divided into two 1 cup daily doses with each of two main meals. After a 3-week washout period, each group will receive the alternative treatment for an additional 2 weeks. Participants will be asked to refrain from making any additional changes to their usual diet throughout the duration of the entire study.

Fasting blood samples will be collected at the beginning and end of each dietary intervention. At the beginning and end of each dietary intervention an additional fasting blood sample will be collected at least one day apart from the main blood collection day for measurement of serum lipids to account for day-to-day variability. Outcome measures include a complete lipid panel (total cholesterol, HDL-c, LDL-c, and triglycerides), fasting glucose, insulin, oxidized LDL and LDL susceptibility to oxidation, total antioxidant capacity (TAC), and vitamin C.

ELIGIBILITY:
Inclusion Criteria:

* Moderate hypercholesterolemia (LDL cholesterol ≥ 120 mg/dL)

Exclusion Criteria:

* Use of hypolipidemic medications
* Regular physical activity (≥ 30 min /day for ≥ 5 days/week)
* Presence of known chronic diseases (e.g., diabetes, CVD, cancer, hepatitis, inflammatory conditions, gastrointestinal disorders)
* Consumption of > 4 servings/day of fruits and vegetables
* Following a restrictive diet (e.g., carbohydrate restriction, veganism) or having any condition likely to require specialized dietary modifications
* Use of supplements (antioxidants, fiber and botanicals)
* Latex allergy
* Fear of needles
* Breastfeeding, pregnancy, or intent to become pregnant
* Unwillingness to comply with study protocol
* Participation in other research studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Plasma lipids | Pre- and post- each 2-week phase
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides.

SECONDARY OUTCOMES:
Glucose | Pre- and post- each 2-week phase
  Plasma glucose
Distribution of cholesterol in LDL and HDL subfractions | After each 2-week phase
  Distribution of cholesterol among seven LDL and ten HDL subfractions.
Oxidized LDL | Pre- and post- each 2-week phase
  Amount of oxidized LDL as measured by ELISA and LDL oxidizability as measured by conjugated diene formation.

OTHER OUTCOMES:
Vitamin C | Pre- and post- each 2-week phase
  Vitamin C concentration in plasma to assess compliance

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Vega-López, PhD, Principal Investigator — Arizona State University
Locations (1):
- Nutrition Laboratory at Arizona State University, Phoenix, Arizona, United States